CLINICAL TRIAL: NCT01700738
Title: Evaluation of the Effects of Laying Early (Between 12 and 16) a Gastric Band on the Prevention of Morbid Obesity in Late Adolescence. Randomized Checked Against Standard Management of Obesity in This Population.
Brief Title: Evaluation of the Effects of Laying Early a Gastric Band on the Prevention of Morbid Obesity Randomized Checked Against Standard Management of Obesity in This Population.
Acronym: CHADO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012 - A00555-38
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gastric ring surgery (Experimental): in this group a gastric ring will be put by surgery.
  Interventions: Procedure: gastric ring surgery
- nutritional help (Active Comparator): the usual treatment of obesity in France with nutritional care will be dispensed for this arm
  Interventions: Other: nutritional help

INTERVENTIONS:
Procedure: gastric ring surgery
  Arms: gastric ring surgery
Other: nutritional help
  Arms: nutritional help

SUMMARY:
MAIN OBJECTIVE To compare the effects of the placement of an adjustable gastric band with "conventional" treatment of obesity.

SECONDARY OBJECTIVES

* Compare the effects of the placement of a gastric band with "conventional" treatment of obesity on quality of life, body composition and parameters of the metabolic syndrome.
* Identify predictors of "good answer to the ring" to determine the best future indications.
* Study of the gastric tolerance.

INCLUSION CRITERIA

1. Adolescents 12 to 16 years and with BMI and weight gain according to sex and age is greater than IMCZ-score > 4 DP> 8 kg
2. Obesity "common" non-syndromic.
3. Medical decision of surgical placement of laparoscopic gastric banding.
4. Adolescent and family who understand and accept the need for medical and surgical follow long term.
5. Adolescent and family who fully understood the oral and written information explaining the study and the need for prolonged follow-up.
6. Obtention of oral and written consent of the adolescent and the parents.
7. Parents and adolescents affiliated with the social security system.

NONINCLUSION CRITERIA

1. Intellectual Deficit.
2. psychiatrics contraindication of surgical placement of laparoscopic gastric banding.
3. Obesity with severe binge eating.
4. Pregnancy or wishes of pregnancy in the following year.
5. Non accession adolescent and / or family in the process of medical care before inclusion.
6. Predictable post surgical monitoring difficulties.
7. Suspicion of physical abuse, verbal or negligence / deficiency in care of the family.
8. Participation in a clinical study evaluating a treatment during the 2 years of the study.

EXCLUSION CRITERIA

1. Anesthetic contre indication for placement of a gastric laparoscopic.
2. IMC> 50 kg/m2 the day of inclusion.

STRATEGIES / PROCEDURES During a routine visit, the study will be presented to the patient and his family. Patients will then be enrolled and randomized. Patients in group A (surgery group) will follow the usual multidisciplinary bariatric surgery in adolescents. Patients in group B start conventional monitoring dietary medical and physical. For both groups follow-up visits will occur every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents 12 to 16 years and with BMI and weight gain according to sex and age is greater than IMCZ-score > 4 DP> 8 kg
2. Obesity "common" non-syndromic.
3. Medical decision of surgical placement of laparoscopic gastric banding.
4. Adolescent and family who understand and accept the need for medical and surgical follow long term.
5. Adolescent and family who fully understood the oral and written information explaining the study and the need for prolonged follow-up.
6. Obtention of oral and written consent of the adolescent and the parents.
7. Parents and adolescents affiliated with the social security system.

EXCLUSION CRITERIA

1. Intellectual Deficit.
2. psychiatrics contraindication of surgical placement of laparoscopic gastric banding.
3. Obesity with severe binge eating.
4. Pregnancy or wishes of pregnancy in the following year.
5. Non accession adolescent and / or family in the process of medical care before inclusion.
6. Predictable post surgical monitoring difficulties.
7. Suspicion of physical abuse, verbal or negligence / deficiency in care of the family.
8. Participation in a clinical study evaluating a treatment during the 2 years of the study.
9. Anesthetic contre indication for placement of a gastric laparoscopic.
10. IMC> 50 kg/m2 the day of inclusion.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
BMIZ-score evolution in 2 years. | 2 years

SECONDARY OUTCOMES:
Evolution of quality of life scales | 1, 2, 5 and 10 years
Evaluation of des alimentary attitudinal troubles and psychiatrical troubles | 1 year
Evolution of BMIZ-score | 1, 5 and 10 years
Evolution of round-waist | 1, 2, 5 and 10 years
Evolution of bodily composition. | 1, 2, 5 and 10 years
Evolution of metabolic syndrome parameters. | 1, 2, 5 and 10 years
Evolution of respiratory parameters: polysomnography | 2 years
Determination of success factors of the ring. | 2 years
Study of tolerance of the gastric ring. | 1, 2, 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: REGIS COUTANT, Principal Investigator — UNIVERSITY HOSPITAL OF ANGERS
Locations (6):
- France (6):
  - University Hospital of Angers, Angers, France
  - University Hospital of Caen, Caen
  - University hospital Bicêtre, Le Kremlin-Bicêtre
  - University Hospital of Lille, Lille
  - University Hospital of Necker, Paris
  - University Hospital of Toulouse, Toulouse

REFERENCES:
- [Derived] Pourcher G, De Filippo G, Ferretti S, Piquard C, Dagher I, Bougneres P. Short-term results of single-port sleeve gastrectomy in adolescents with severe obesity. Surg Obes Relat Dis. 2015 Jan-Feb;11(1):65-9. doi: 10.1016/j.soard.2014.05.029. Epub 2014 Jun 3. PMID 25393047